CLINICAL TRIAL: NCT02210624
Title: An Open-label, Safety and Efficacy Assessment of Autologous Bone-marrow Derived Mesenchymal Stem Cell Therapy in Anoxic (or Hypoxic) Brain Injury.
Brief Title: Safety and Efficacy Assessment of Autologous Bone-marrow Derived Adult Mesenchymal Stem Cell Therapy in Patients With Anoxic(or Hypoxic) Brain Injury Pilot Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hyun Young Kim (Other)
Responsible Party: Sponsor-Investigator, Hyun Young Kim, seong joon kwon, Hanyang University Seoul Hospital
Organization: Hanyang University Seoul Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYNR_CS_ABI001
Record Dates: First submitted 2014-07-31; First posted 2014-08-07 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Anoxic Brain Injury
Keywords: Anoxic Brain Injury; Autologous bone marrow derived stem cell; stoke
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Experimental: HYNR-CS inj.
  Treatment group with HYNR-CS inj.
  Interventions: Biological: HYNR-CS inj.

INTERVENTIONS:
Biological: HYNR-CS inj. — Intrathecal injection with 1ml/10kg of body weight at an interval of 26 days.

SUMMARY:
The purpose of study is to evaluate the safety and efficacy of autologous bone marrow-derived stem cells therapy in patients with anaerobic (hypoxic) brain injury. Stem cell therapy is an emerging alternative treatment modality in incurable and intractable neurological disorders. This pilot study aims to evaluate the feasibility and safety of stem cells in anaerobic brain injury.

DETAILED DESCRIPTION:
Various treatment modalities to minimize the neurological deficits of anoxic brain injury, including lower consciousness, abnormal movement disorders, and abnormal behavior, have been tried, but so far there have been no effective proven method for chronic patients.

This study is the investigator initiated trial to verify the safety and feasibility of stem cells therapy in patients with anoxic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 14 days after the index event occurs in an oxygen-free brain injury patients
* Severe disability or moderate due to anoxic brain injury
* 18 years to 75 years
* Patients was 7 points less than Glasgow coma scale (GCS) After the resumption of blood flow circulation.
* anaerobic unexpected (hypoxic) cerebral ischemia Encephalopathy (It should not be a hypoxic brain ischemia was induced due to heart surgery, which is scheduled)
* Subjects agreed in writing that it will be participating in clinical research, as viewed from the legal representative (patient)

Exclusion Criteria:

* Patients who require ventilator continued
* Patients who had extracorporeal membrane oxygenation(ECMO) index event occurs at the time
* Patients who had a history of cardiac arrest prior to the occurrence of Index event
* End-stage people of less than 12 months is expected (incurable) disease patients
* Patients with cardiac arrest occurred due to brain trauma severe
* Patients with damage to other organs of severe
* Patients with bleeding or malignant current
* Pregnant patient
* Patients with central nervous system tumors undergoing radiation therapy or chemotherapy
* If the patient or are participating in other clinical trials, you are planning to participate, or patients three months after the end is not passed to participate in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
safety assessment | week 1, 3, 4, 5, 7
  Each visit physical examination, neurological examination, and adverse reactions through the follow-up to the expression of new symptoms.
  week 1,3,5,7 conducted Hematological week 4,7 conducted MRI, PET

SECONDARY OUTCOMES:
Glasgow Coma Scale(GCS) | Week 1, 4, 5, 6, 7
  assess level of consciousness after head injury
FOUR score | Week 1, 4, 5, 6, 7
  The FOUR Score is a clinical grading scale designed for use by medical professionals in the assessment of patients with impaired level of consciousness.
Functional Independence Measure(FIM) | Week 1, 4, 5, 6, 7
  The Functional Independence Measure (FIM™) instrument is a basic indicator of patient disability.
Disability Rating Scale(DRS) | Week 1, 4, 5, 6, 7
  The Disability Rating Scale (DRS) is primarily used to assess impairment, disability, and handicap of an individual.
Cerebral Performance Category(CPC)scale | Week 1, 4, 5, 6, 7
  The Cerebral Performance Category score is to use measure of functional outcome after cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Young Kim, MD.,PhD., Principal Investigator — Hanyang University
Locations (1):
- Hanyang University Hospital, Seoul, South Korea